CLINICAL TRIAL: NCT06628336
Title: Post-Market Observational Study of the HARMONY® Evolution Implants and Instruments
Status: Recruiting | Type: Observational
Sponsor: Symbios Orthopedie SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-H-035
Record Dates: First submitted 2024-05-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Total Hip Replacement
Keywords: HARMONY; THR; Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HARMONY EVOLUTION — It is planned to include consecutive eligible subjects which will be treated with the HARMONY EVOLUTION devices.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the HARMONY® Evolution implants in a series of operated subjects treated in THR.

The objective is to demonstrate that the evaluated implants are compliant with the state of the art and the performance (PMA score > 15 points) & safety claims (The expected acceptable revision rate (state of the art with a confidence interval of 95%) is 3% at 3 years, 5% at 5 years, 7% at 7 years and 10% at 10 years).

The endpoint of this study is to validate the expected performance of the HARMONY® Evolution implants with the PMA score at 10 years and to validate the safety claim with the expected acceptable revision rate at 10 years.

DETAILED DESCRIPTION:
The study is prospective, multi-centric, observational, non-comparative, non-randomized and post market. About 264 subjects will be enrolled in this study to evaluate the safety and performance of the HARMONY® Evolution implants.

Patients will be included in the study during 12 months and followed-up during 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 18 years of age and older
* Each subject who is willing to give informed consent
* Clinically indicated for a Total Hip Replacement
* Women of childbearing age who are not pregnant and do not expect to become pregnant within 12 months. A pregnancy test should be performed for women of childbearing age
* Geographically stable and willing to return to the implanting site for all follow-up visits

Exclusion Criteria:

* Acute or chronic, local or systemic infection
* Muscular, neurological, psychological or vascular deficits
* Poor bone density and quality likely to affect implant stability (severe osteoporosis)
* Any concomitant condition likely to affect implant integration or function
* Allergy or hypersensitivity to any of the materials used

Specific:

• The HARMONY® Evolution Standard stem size 8 shall not be implanted in subjects weighing more than 70 kg.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have provided consent for the collection of their data and met the protocol eligibility criteria will be enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2034-10-11 (Estimated); Study Completion 2035-03-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety by means of measuring Adverse event recurrences | 2 months, 1, 3, 5 and 10 years follow-up
  Proportion of patients requiring a revision.
Evaluate performance by means of clinical and quality of life scores | 2 months, 1, 3, 5 and 10 years follow-up
  Score PMA > 15 points

SECONDARY OUTCOMES:
Evaluate performance by means of surgeon satisfaction questionnaire | 2 months, 1, 3, 5 and 10 years follow-up
  Evaluate the success of the surgical procedure and evaluate surgeon satisfaction regarding the implant components and the use of instruments with the criteria: very satisfied - satisfied - unsatisfied - very unsatisfied for each surgical step.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Castelain, Dr., Principal Investigator — Clinique Arago
Locations (5):
- France (5):
  - Polyclinique de Franche-Comté, Besançon
  - Clinique Belledonne, Grenoble
  - Clinique Juge, Marseille
  - Clinique Arago, Paris
  - Médipôle Garonne, Toulouse

IPD SHARING:
Plan to Share IPD: No